CLINICAL TRIAL: NCT00929760
Title: Impact of Specialised Renal Care in Patients With Chronic Kidney Disease Stage 3-5: A Prospective Randomised Study. "The Implicate Study"
Brief Title: Impact of Specialised Renal Care in Patients With Chronic Kidney Disease
Acronym: IMPLICATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patrick Saudan (Other)
Collaborators: Schweizerische Nierenliga (Unknown)
Responsible Party: Sponsor-Investigator, Patrick Saudan, Professor, MD, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-226
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2009-09

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney disease; Nephrologists; Primary Care; Death; Renal Replacement Therapy; Specialised renal care
MeSH Terms: conditions — Renal Insufficiency, Chronic; Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nephrologists (Active Comparator): Combined management PCP: nephrologists (at least 4 nephrology visits/year)
  Interventions: Behavioral: specialised renal care
- Primary Care Physicians (Active Comparator): Management by PCPs only, with the help of written instructions from our nephrology unit based on EBPG
  Interventions: Behavioral: specialised renal care

INTERVENTIONS:
Behavioral: specialised renal care — * Combined management PCP - nephrologists (at least 4 nephrology visits/year). Agreement of the PCP is required for this combined management.
  * Management by PCPs only, with the help of written instructions from our nephrology unit based on EBPG. Requested Email or over the phone advices to PCPs will be provided by the nephrology division of HUG.

SUMMARY:
This is a prospective randomised trial studying patients with stage 3 to 5 chronic kidney disease (CKD) in order to determine the impact of specialised care by nephrologists compared to guidelines-directed management by primary care physicians (PCP) on: a) prognosis (clinical outcome), b) planning of renal replacement therapy (RRT) (urgent versus planned initiation RRT) and c) patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD stage 3, 4 and 5 (CCl < 40 ml/min according to abbreviated MDRD formula) aged 18-80 years old and enrolled during a hospitalization.

Exclusion Criteria:

* Patients previously known by nephrologists.
* Estimated life expectancy < 1 year
* Refusal or inability to sign writing consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2009-06; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Primary (composite): death, and hospitalisation | 24 months after enrollment
  death and emergency hospitalisation during the following 2 years afterr andomisation

SECONDARY OUTCOMES:
Secondary: initiation of urgent RRT, decline of renal residual function at 2 years, decline of quality of life | 24 months after enrollment
  cf title

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Unit Geneva University Hospitals, Geneva, Geneva City, Switzerland

REFERENCES:
- [Derived] Saudan P, Ponte B, Marangon N, Martinez C, Berchtold L, Jaques D, Ernandez T, de Seigneux S, Carballo S, Perneger T, Martin PY. Impact of superimposed nephrological care to guidelines-directed management by primary care physicians of patients with stable chronic kidney disease: a randomized controlled trial. BMC Nephrol. 2020 Apr 9;21(1):128. doi: 10.1186/s12882-020-01747-3. PMID 32272886